CLINICAL TRIAL: NCT02647918
Title: A Phase 1, Open-label, Parallel-group Study to Evaluate Sotagliflozin Safety and Pharmacokinetics in Subjects With Varying Degrees of Renal Function
Brief Title: Study to Evaluate Sotagliflozin in Subjects With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-121-REN; LX4211.121 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Renal Impairment; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Subjects with normal renal function
  Interventions: Drug: Sotagliflozin
- Group 2 (Experimental): Subjects with mild renal impairment
  Interventions: Drug: Sotagliflozin
- Group 3 (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: Sotagliflozin
- Group 4 (Experimental): Subjects with severe renal impairment
  Interventions: Drug: Sotagliflozin
- Group 5 (Experimental): Subjects with ESRD requiring HD
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Single dose
  Arms: Group 1; Group 2; Group 3; Group 4
Drug: Sotagliflozin — 2 single doses
  Arms: Group 5

SUMMARY:
The purpose of this study is to evaluate the effect of mild, moderate, or severe renal impairment, or end-stage renal disease (ESRD) requiring hemodialysis (HD), on the safety and tolerability of 1 or 2 single doses of sotagliflozin compared with healthy, demographically-matched subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects ≥18 to ≤75 years of age
* Body mass index ≥18.0 to ≤36.0 kg/m2, at Screening
* Subjects with mild, moderate, or severe renal impairment, or ESRD requiring HD
* Control group of matched healthy subjects
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings that may interfere with any aspect of study conduct or interpretation of results
* Existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism, or excretion of sotagliflozin
* History of any major surgery within 6 months
* History of hepatic disease, or significantly abnormal liver function test
* Women who are breastfeeding or are planning to become pregnant during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | Day 1 to Day 8

SECONDARY OUTCOMES:
Plasma concentration of sotaglifozin to evaluate AUC | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Minneapolis, Minnesota
  - Lexicon Investigational Site, Saint Paul, Minnesota